CLINICAL TRIAL: NCT04092907
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled Study Evaluating the Efficacy and Safety of HBM9036 Ophthalmic Solution Versus Placebo in Subjects With Moderate to Severe Dry Eye
Brief Title: A Study Evaluating the Efficacy and Safety on Moderate to Severe Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9036.1
Record Dates: First submitted 2019-09-09; First posted 2019-09-17 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBM9036 0.25% Ophthalmic Solution (Experimental): HBM9036, Ophthalmic Solution, twice a day, in the morning and evening
  Interventions: Drug: HBM9036 0.25% Ophthalmic Solution
- Placebo Ophthalmic Solution (Placebo Comparator): placebo, Ophthalmic Solution, twice a day, in the morning and evening
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HBM9036 0.25% Ophthalmic Solution — Ophthalmic Solution
  Arms: HBM9036 0.25% Ophthalmic Solution
Drug: placebo — Ophthalmic Solution
  Arms: Placebo Ophthalmic Solution

SUMMARY:
The purpose of this study is to compare the efficacy and safety of HBM9036 Ophthalmic Solution versus placebo in the treatment of dry eye

DETAILED DESCRIPTION:
HBM9036 is a molecularly engineered tumor necrosis factor receptor 1 (TNFR1) fragment.

A total of 100 subjects are expected to be randomized. Subjects will be randomized 1:1 at Visit 2 to HBM9036 Ophthalmic Solution or placebo group, bilaterally BID for eight weeks. The primary efficacy endpoint is sign changes from baseline in change from pre- to post-CAE inferior corneal staining score (ICSS) of the study eye evaluated at week 8 .

ELIGIBILITY:
Inclusion Criteria

1. Have a history of use eye drops for dry eye symptoms within 6 months of Visit 1 or desire to use eye drops;
2. Have in the study eye a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm at Visits 1 and 2;
3. Be willing and can adjust current treatment for dry eye according to the protocol, judged by the Investigator;
4. Must be willing to complete all study assessments required by the protocol.

Exclusion Criteria:

1. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
2. Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months, or had femtosecond small incision lenticule extraction (SMILE) within the last 12 months, or had phacoemulsification within the last 3 months, or had dry eye or aggravation of dry eye caused by other ocular operations has not been stable;
3. Have used ophthalmic cyclosporine A, tacrolimus or Xiidra® within 60 days prior to Visit 1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lixin XIE, Academician, Principal Investigator — QINGDAO EYE HOSPITAL
Locations (1):
- Qingdao Eye Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong Y, Wang S, Cong L, Zhang T, Cheng J, Yang N, Qu X, Li D, Zhou X, Wang H, Lee M, Wang M, Chen S, Ousler GW, Chen X, Xie L. TNF-alpha inhibitor tanfanercept (HBM9036) improves signs and symptoms of dry eye in a phase 2 trial in the controlled adverse environment in China. Int Ophthalmol. 2022 Aug;42(8):2459-2472. doi: 10.1007/s10792-022-02245-1. Epub 2022 Feb 22. PMID 35192105

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HBM9036 0.25% Ophthalmic Solution | Placebo Ophthalmic Solution
Started | 50 | 50
Completed | 48 | 50
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants screened for whom a randomization number was assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | HBM9036 0.25% Ophthalmic Solution | Placebo Ophthalmic Solution | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.19) | 43.9 (9.15) | 42.6 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 25 | 18 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Inferior Corneal Staining (ICS) Score
Description: Inferior corneal staining score, assessed by Ora Calibra® Corneal and Conjunctival Fluorescein Staining Scale (0-4 point, higher is worse) Change from baseline in change from pre- to post- CAE at Visit 6 (higher is worse)
Time Frame: 8 weeks
Population: The analysis population is per-protocol population, which excluded a few patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HBM9036 0.25% Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 47 | 48
units on a scale | 1.8 (0.44) | 1.9 (0.46)

2. Secondary Outcome: Ocular Discomfort Score
Description: Ocular Discomfort Score, assessed by Ora Calibra® Ocular Discomfort Scale (0-4 point, higher is worse) Change from baseline in pre-CAE Ocular Discomfort Score at Visit 6 (higher is worse)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HBM9036 0.25% Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 47 | 48
units on a scale | 2.94 (0.791) | 3.10 (0.692)

ADVERSE EVENTS:
Time Frame: From start of the first study drug administration up to Day 57 or Early termination (ET)
Description: Adverse events that occurred after the start of first dose administration are considered treatment emergent adverse and summarized by treatment arm. A participant (subject) is counted only once for the same adverse event, regardless of the number of episodes.
Arm/Group | HBM9036 0.25% Ophthalmic Solution | Placebo Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 14/50 | 14/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HBM9036 0.25% Ophthalmic Solution (N=50) | Placebo Ophthalmic Solution (N=50)
Conjunctival hyperemia (Eye disorders) | 3 | 0
Eye pruritus (Eye disorders) | 1 | 1
Allergic conjunctivitis (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Ocular pain (Eye disorders) | 1 | 0
Visual fatigue (Eye disorders) | 1 | 0
Ocular hyperemia (Eye disorders) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 3 | 0
Subepidermal hemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 5
Local infection (Infections and infestations) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
rhinobyon (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mouth ulcers (Gastrointestinal disorders) | 1 | 0
toothache (Gastrointestinal disorders) | 0 | 1
gastritis (Gastrointestinal disorders) | 0 | 1
backache (Musculoskeletal and connective tissue disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Skin trauma (Injury, poisoning and procedural complications) | 0 | 1
Sprained ligament (Injury, poisoning and procedural complications) | 0 | 1
Seasonal allergies (Immune system disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04092907/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04092907/SAP_001.pdf
  • Informed Consent Form (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04092907/ICF_002.pdf